CLINICAL TRIAL: NCT01252017
Title: Cytomegalovirus (CMV) Reactivation in Post-allogeneic Hematopoietic Stem Cell Transplantation(Allo-HSCT) Patients: Salvage and Prophylactic Treatments of Nilotinib
Brief Title: Nilotinib for Cytomegalovirus Prophylaxis and Treatment After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201006057M
Record Dates: First submitted 2010-11-24; First posted 2010-12-02 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Patients Who Have Received Allo-HSCT
MeSH Terms: interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental): Single arm, open label study
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — nilotinib (200mg/tab) 1 tab everyday
  Other Names: tasigna

SUMMARY:
The purpose of this study is to determine whether nilotinib is effective in the prophylaxis and treatment of CMV reactivation in allo-HSCT patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether nilotinib is effective in the prophylaxis and treatment of CMV reactivation in allo-HSCT patients.

Prophylaxis Part: patients will be treated with nilotinib after their hemogram engraftment to prevent CMV reactivation Salvage Part: patients who have had intractable CMV reactivation after gancyclovir therapy will be treated with nilotinib

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Adult patients who have received allo-HSCT
* Performance status ECOG 0-2
* Patients with CMV reactivation (defined as plasma CMV DNA copy numbers of more than 1000 copy numbers/ml by Quantitative-PCR) after allo-HSCT.
* Patients with CMV reactivation that is uncontrollable by conventional first line agent (ganciclovir) for 2 or more weeks, or patients who are intolerable to ganciclovir treatment.

Part B

* Adult patients who have received allo-HSCT
* Performance status ECOG 0-2
* Either the patient or his/her donor are CMV-IgG test positive
* Patients with post-transplantation engraftment: stable myeloid engraftment (absolute neutrophil count 500/mm3) for at least 3 consecutive days, and stable megakaryocyte engraftment (platelet count 20k/uL) for at least 3 consecutive days.
* Patient with no CMV reactivation before enrollment: a negative (undetectable) plasma CMV DNA Quantitative-PCR assay on blood collected within 7 days Patients without previous or current exposure to any prophylactic or therapeutic drugs for CMV reactivation

Exclusion Criteria:

* Patients with renal insufficiency: serum creatinine > 2.5 mg/dL,
* Patients with significant electrolyte deficiency after suitable supplement: [K] <3.0mmol/L, [Ca]< 2.0 mmol/L(corrected), or [Mg] < 0.6 mmol/L.
* Patients with hepatic dysfunction: alkaline phosphatase ≥2.5 times of the upper normal limit of the normal range (ULN); serum alanine or aspartate aminotransferase levels of > 5 times ULN; a serum total bilirubin of > 3 mg/dL
* Patients with serum amylase and lipase > 1.5 x ULN
* Patients with history of HIV infection
* Patients with unstable medical condition or any other history of serious/significant medical diseases deemed not appropriate to be included to this study as judged by investigators
* Females patient who are pregnant or breast-feeding
* Female patients of childbearing potential not using any reliable and appropriate contraception method(s)
* Patients with life expectancy, as judged by the investigators, is less than 3 months
* Patients with, as judged by the investigators, other contraindications of nilotinib administration, such as prolonged QTc, concurrent usage of drugs that possess possible severe drug-drug interactions with nilotinib, or had severe adverse effects in the previous exposure to nilotinib
* Patients who cannot swallow capsules.
* Patients who are unwilling or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
anti-CMV treatment free rate | 100 days after allo-HSCT (Day+100)
  For prophylaxis part

SECONDARY OUTCOMES:
Successful salvage rate | up to 8 weeks
  For salvage treatment part

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Ju Wu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Lin CT, Hsueh PR, Wu SJ, Yao M, Ko BS, Li CC, Hsu CA, Tang JL, Tien HF. Repurposing Nilotinib for Cytomegalovirus Infection Prophylaxis after Allogeneic Hematopoietic Stem Cell Transplantation: A Single-Arm, Phase II Trial. Biol Blood Marrow Transplant. 2018 Nov;24(11):2310-2315. doi: 10.1016/j.bbmt.2018.07.013. Epub 2018 Jul 17. PMID 30026110